CLINICAL TRIAL: NCT07382349
Title: Randomized Controlled Trial of Electronic Clinical Decision Support Systems for Improving Care Management and Clinical Outcomes for Adults With Steatotic Liver Disease
Brief Title: A Study of Electronic Clinical Decision Support Tools for Steatotic Liver Disease
Acronym: eMPOWER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: American Association for the Study of Liver Diseases (Other)
Responsible Party: Principal Investigator, Ashley Spann, Assistant Professor, Transplant Hepatology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 241192
Record Dates: First submitted 2026-01-24; First posted 2026-02-02 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: MASLD
Keywords: Electronic Health Record; MASLD; Clinical Decision Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Group (No Intervention): Care providers will treat subject per standard of care
- Electronic Decision Aid Group (Experimental): the eMPOWER Decision Aid will be used to alert care providers to the patient specific recommendations for management of steatotic liver disease based on risk stratification
  Interventions: Other: eMPOWER Decision Aid

INTERVENTIONS:
Other: eMPOWER Decision Aid — An electronic health record embedded decision aid utilizing clinical data from both structured and unstructured clinical data to guide risk stratification and care management for patients with steatotic liver disease. Providers will be alerted to patient specific recommendations during the clinical encounter and between encounters through asynchronous communications related to subsequent testing.
  Arms: Electronic Decision Aid Group

SUMMARY:
The overall objectives of this study are to determine the effectiveness of a participant-specific guided electronic decision support system on provider decision making for participants with metabolic-dysfunction associated steatotic liver disease (MASLD), and to determine the acceptance and barriers for use of an electronic health record embedded algorithm for MASLD care management within ambulatory primary care, endocrinology, and general gastroenterology settings.

DETAILED DESCRIPTION:
A pragmatic, randomized trial within selected clinical practices for primary care, endocrinology, and non-hepatology gastroenterology sites within Vanderbilt University Medical Center will be conducted over a period of 3 years with 12 months of follow up for each participant. Participants will be randomized 1:1 to intervention or usual care. In the intervention arm, the decision support aid (eMPOWER) will be used to alert consenting providers to participant-specific recommendations for steatotic liver disease care based on clinical features and risk factor profiles. The primary endpoint will be linkage to care determined by orders for referral to hepatology for advanced liver disease. Secondary outcomes will include completion of noninvasive fibrosis assessment tests for indeterminate risk participants by FIB-4 (1.3-2.67 for participants under 65, 2.0-2.67 for participants 65 and older), completion rates of hepatology referrals, and time analyses to complete either referrals or elastography studies. Post-study surveys and interviews to participating clinicians will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 years)
* Outpatient clinic visit (in-person or telemedicine) at a participating clinic site
* Demonstrated Screening Need due to High Risk Profile, which includes the following: Diagnostic Codes for MASLD or Hepatic Steatosis on Imaging PLUS at least one cardiometabolic risk factors; OR Chronically Elevated Liver Enzymes (> 6 months); OR patient with impaired glycemic control (prediabetes/diabetes); OR 2 or more cardiometabolic risk factors present

Exclusion Criteria:

* Solid Organ Transplant Recipient
* Existing Hepatology Relationship Evidenced by Prior Hepatology Visit Within 3 Years
* Active Cancer Diagnoses
* Diagnoses for Alcohol-Related Conditions
* Pregnant Individuals
* Receiving Palliative Care Services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7200 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this pragmatic trial is to assess the efficacy of the electronic decision support aid for increasing linkage to hepatology care for high-risk participants with MASLD | Baseline to 12 months
  Number of participants with new referrals placed to Hepatology for evaluation of high-risk status

SECONDARY OUTCOMES:
The secondary objective is to assess the efficacy of the electronic decision support aid for increasing elastography testing ordered by primary care and specialty care providers for indeterminate-risk participants with MASLD | Baseline to 12 months
  Number of participants with orders placed by primary care and specialty care providers for noninvasive elastography assessments for evaluation of indeterminate risk status
Rate of Completion of Hepatology Referral | Baseline to 12 months
  Of patients referred to Hepatology, number of participants with completed referrals for evaluation of high-risk status
Time to Completion of Hepatology Referral | Baseline to 12 months
  Of patients referred to Hepatology, time to completion of referrals placed to Hepatology for evaluation of high-risk status determined by FIB-4 scoring
Rate of Completion of Noninvasive Elastography Studies | Baseline to 12 months
  Of patients ordered for noninvasive fibrosis testing, number of completed orders placed by primary care and specialty care providers for evaluation of indeterminate risk status
Time to Completion of Noninvasive Elastography Studies | Baseline to 12 months
  Of patients ordered for noninvasive fibrosis testing, time to completion of orders placed by primary care and specialty care providers for evaluation of indeterminate risk status

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Spann, MD, MSACI, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
Protected Health Information

REFERENCES:
- [Background] Spann A, Bishop KM, Weitkamp AO, Stenner SP, Nelson SD, Izzy M. Clinical decision support automates care gap detection among primary care patients with nonalcoholic fatty liver disease. Hepatol Commun. 2023 Feb 9;7(3):e0035. doi: 10.1097/HC9.0000000000000035. eCollection 2023 Mar 1. PMID 36757410
- [Background] Spann A, Bishop K, Marbach S, Ji X, Slaughter J, Weitkamp A, Stenner S, Nelson S, Lopez C, Theobald C, Izzy M. Electronic decision aids enhance management of primary care patients with steatotic liver disease: Proof of concept pilot study. Hepatol Commun. 2025 Sep 5;9(9):e0794. doi: 10.1097/HC9.0000000000000794. eCollection 2025 Sep 1. PMID 40906885